CLINICAL TRIAL: NCT01034267
Title: A Long-Term, Open-label Extension Study of F2695 SR in Adult Patients With Major Depressive Disorder
Brief Title: Safety Study of F2695 SR in Major Depressive Disorder
Acronym: LVM-MD-04
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LVM-MD-04
Record Dates: First submitted 2009-12-16; First posted 2009-12-17 (Estimated); Last update posted 2012-08-17 (Estimated); Status verified 2012-08

CONDITIONS: Major Depressive Disorder
Keywords: Depression; Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): (Open-label) F2695 SR capsules, oral administration, once daily, flexible dosing
  Interventions: Drug: F2695 SR

INTERVENTIONS:
Drug: F2695 SR — Drug F2695 SR (flexible dose) to be given orally in capsule form once daily

SUMMARY:
The purpose of this study is to evaluate the long- term safety of F2695-SR in the treatment of adults with major depressive disorder.

ELIGIBILITY:
Inclusion Criteria:

* Completed 1 of the lead-in studies LVM-MD-01, LVM-MD-02, or LVM-MD-03
* Have normal examination findings at the final visit of the lead-in study
* Have a negative serum pregnancy test at the final visit of the lead-in study if a woman of child-bearing potential

Exclusion Criteria:

* Any exclusionary psychiatric or medical condition that developed during the lead in study
* Patients considered a suicide risk
* Women who are pregnant, breastfeeding, or planning to become during the study OR are sexually active and not currently using a medically acceptable method of contraception

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 828 (Actual)
Dates: Start 2009-12; Primary Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Adverse events, clinical laboratory tests, vital sign measurements, electrocardiograms, physical examinations, Columbia-Suicide Severity Rating Scale | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Giovana Forrero, MA, Study Director — Forest Research Institute, a subsidiary of Forest Laboratories Inc
Locations (68):
- United States (68):
  - Forest Investigative Site 55, Dothan, Alabama
  - Forest Investigative Site 29, Scottsdale, Arizona
  - Forest Investigative Site 31, Beverly Hills, California
  - Forest Investigative Site 3, Costa Mesa, California
  - Forest Investigative Site 12, Encino, California
  - Forest Investigative Site 6, Escondido, California
  - Forest Investigative Site 22, Oceanside, California
  - Forest Investigative Site 38, Sherman Oaks, California
  - Forest Investigative Site 36, Denver, Colorado
  - Forest Investigative Site 28, Denver, Colorado
  - Forest Investigative Site 65, Highlands Ranch, Colorado
  - Forest Investigative Site 30, Cromwell, Connecticut
  - Forest Investigative Site 57, Boca Raton, Florida
  - Forest Investigative Site 60, Boca Raton, Florida
  - Forest Investigative Site 18, Coral Springs, Florida
  - Forest Investigative Site 34, Fort Myers, Florida
  - Forest Investigative Site 64, Gainesville, Florida
  - Forest Investigative Site 45, Hallandale, Florida
  - Forest Investigative Site 17, Jacksonville, Florida
  - Forest Investigative Site 53, Ocala, Florida
  - Forest Investigative Site 13, Orlando, Florida
  - Forest Investigative Site 61, Orlando, Florida
  - Forest Investigative Site 27, West Palm Beach, Florida
  - Forest Investigative Site 59, Winter Park, Florida
  - Forest Investigative Site 70, Atlanta, Georgia
  - Forest Investigative Site 66, Smyrna, Georgia
  - Forest Investigative Site 33, Chicago, Illinois
  - Forest Investigative Site 23, Hoffman Estates, Illinois
  - Forest Investigative Site 50, Oak Brook, Illinois
  - Forest Investigative Site 63, Indianapolis, Indiana
  - Forest Investigative Site 71, Prairie Village, Kansas
  - Forest Investigative Site 5, Wichita, Kansas
  - Forest Investigative Site 52, Shreveport, Louisiana
  - Forest Investigative Site 1, Baltimore, Maryland
  - Forest Investigative Site 2, Glen Burnie, Maryland
  - Forest Investigative Site 37, Rockville, Maryland
  - Forest Investigative Site 32, Fall River, Massachusetts
  - Forest Investigative Site 15, East Lansing, Michigan
  - Forest Investigative Site 35, Cherry Hill, New Jersey
  - Forest Investigative Site 21, Willingboro, New Jersey
  - Forest Investigative Site 51, Brooklyn, New York
  - Forest Investigative Site 42, Brooklyn, New York
  - Forest Investigative Site 4, Mount Kisco, New York
  - Forest Investigative Site 16, New York, New York
  - Forest Investigative Site 39, New York, New York
  - Forest Investigative Site 9, Staten Island, New York
  - Forest Investigative Site 46, Raleigh, North Carolina
  - Forest Investigative Site 25, Canton, Ohio
  - Forest Investigative Site 10, Dayton, Ohio
  - Forest Investigative Site 56, Oklahoma City, Oklahoma
  - Forest Investigative Site 67, Oklahoma City, Oklahoma
  - Forest Investigative Site 40, Portland, Oregon
  - Forest Investigative Site 58, Salem, Oregon
  - Forest Investigative Site 54, Allentown, Pennsylvania
  - Forest Investigative Site 14, Media, Pennsylvania
  - Forest Investigative Site 43, Norristown, Pennsylvania
  - Forest Investigative Site 24, Philadelphia, Pennsylvania
  - Forest Investigative Site 44, Lincoln, Rhode Island
  - Forest Investigative Site 26, Memphis, Tennessee
  - Forest Investigative Site 20, Dallas, Texas
  - Forest Investigative Site 47, Dallas, Texas
  - Forest Investigative Site 62, San Antonio, Texas
  - Forest Investigative Site 7, San Antonio, Texas
  - Forest Investigative Site 8, Woodstock, Vermont
  - Forest Investigative Site 68, Virginia Beach, Virginia
  - Forest Investigative Site 19, Bellevue, Washington
  - Forest Investigative Site 41, Seattle, Washington
  - Forest Investigative Site 69, Spokane, Washington